CLINICAL TRIAL: NCT02916745
Title: Multicenter, Prospective, OL, Single-arm Clinical Study of Safety & Feasibility of Using Navigational Bronchoscopy to Perform Interstitial PD Therapy Using Photofrin® as Treatment in Subjects With Unresectable Solid Tumor in Peripheral Lung
Brief Title: Feasibility Study of Using Navigational Bronchoscopy to Perform PDT-Photofrin® in Unresectable Peripheral Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concordia Laboratories Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLI-PHO1601
Record Dates: First submitted 2016-09-26; First posted 2016-09-27 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Non-small Cell Lung Cancer (NSCLC); Lung Metastasis
Keywords: Non-small cell lung cancer; NSCLC; lung cancer; lung carcinoma; lung metastasis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Dihematoporphyrin Ether; Optical Fibers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Photodynamic therapy-Photofrin (Experimental): Photodynamic therapy (PDT) involves the i.v. injection of 2 mg/kg-porfimer sodium (Photofrin®) followed by illumination of the tumor using a fiber optic device during navigational bronchoscopy. Two days after the injection, a laser light will be applied to the tumor.
  Interventions: Drug: Porfimer sodium; Device: Fiber optic

INTERVENTIONS:
Drug: Porfimer sodium — After injection of porfimer sodium (Photofrin®), a flexible bronchoscopy with navigation guidance will be performed to confirm the location and the size of the lesion with the use of radial probe endobronchial ultrasonography (REBUS). A light dose of 200 J/cm of diffuser length will be delivered.
  Other Names: Photofrin
Device: Fiber optic — A fiber optic diffuser length matching the tumor length will be placed in the lesion under fluoroscopy guidance.

SUMMARY:
This research study is being conducted to assess the safety and feasibility of using a new developed bronchoscopic technology called electronavigational bronchoscopy to treat subjects with solid tumor in peripheral lung, who are inoperable or refused surgery. It will involve 10 sites in USA and Canada. Participation will last 6 months.

DETAILED DESCRIPTION:
Lung cancer accounts for almost one-third of cancer deaths. Cancer screening strategies have the potential to achieve a 20% reduction in death rates. Newly developed bronchoscopic technologies (such as navigational bronchoscopy) have shown to enable physicians to safely reach lesions in peripheral regions of the lung and obtain diagnosis. This new technology may now potentially offer bronchoscopic therapeutic interventions, such as photodynamic therapy, to tumors that were previously unreachable due to their peripheral anatomic location.

Photodynamic therapy (PDT) uses a combination of a photosensitizing drug (a drug that is activated by light), called porfimer sodium (Photofrin®), and a light from a laser that emits no heat. This technique works to allow the medical doctor to specifically target and destroy abnormal or cancer cells while limiting damage to surrounding healthy tissue. The activation of the drug is done by lighting the abnormal area using a fiber optic device (very fine fiber [like a fishing line] that permits light transmission) inserted into a flexible tube called bronchoscope. The light activates the porfimer sodium, which is concentrated in the abnormal tissue, leading to its destruction.

The purpose of this study is to determine if physicians can reach the tumors in the periphery of the lung via electronavigational bronchoscopy and deliver the photodynamic therapy by placing the optical fiber into the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 or older
* Diagnosed with histologically confirmed solid tumor located in the peripheral lung
* Not candidate for curative surgery, is unfit for surgery, or does not wish to undergo curative surgery
* May be candidate for, have failed, or does not wish to undergo radiation therapy
* The tumor is ≤ 3 cm in size and clearly observable in computerized tomography (CT scan)
* Able to sign an informed consent

Exclusion Criteria:

* Diagnostic of small cell lung cancer
* Solid tumor located in central lung
* Presence of concurrent non-solid malignancy
* Abnormal blood results
* Received chemotherapy/immunotherapy in the last 4 weeks
* Tumor invades a major blood vessel
* Porphyria or known hypersensitivity to Photofrin® or porphyrin-like compounds or to any of its excipients
* Planned surgical procedure within the next 90 days
* Coexisting ophthalmic disease likely to require slit-lamp examination within the next 90 days
* Acute or chronic medical or psychological illnesses that prevent endoscopy procedures
* Pregnant or intend to become pregnant, breastfeeding or intend to breastfeed during the study
* Received PDT during the past 3 months
* Severe impairment of your kidney or liver function
* Participates or intends to participate in another drug study (other than observational studies) during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Depot, Ph.D., Study Director — at the request of Concordia Laboratories Inc.
Locations (7):
- United States (6):
  - University of Florida, Gainesville, Florida
  - Southeastern Regional Medical Center, Atlanta, Georgia
  - Alexian Brothers Hospital Network, Elk Grove Village, Illinois
  - Southwestern Regional Medical Center, Tulsa, Oklahoma
  - Providence Medical Research Center, Spokane, Washington
  - University of Wisconsin-Madison, Madison, Wisconsin
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Photodynamic Therapy-Photofrin
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Photodynamic Therapy-Photofrin: Photodynamic therapy (PDT) involves the intravenous injection of 2 mg/kg-porfimer sodium (Photofrin®) followed by illumination of the tumor using a fiber optic device during navigational bronchoscopy. Two days after the injection, a laser light will be applied to the tumor.
  Porfimer sodium: After injection of porfimer sodium (Photofrin®), a flexible bronchoscopy with navigation guidance will be performed to confirm the location and the size of the lesion with the use of radial probe endobronchial ultrasonography (REBUS). A light dose of 200 J/cm of diffuser length will be delivered.
  Fiber optic: A fiber optic diffuser length matching the tumor length will be placed in the lesion under fluoroscopy guidance.
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.75 (6.99)
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.75 (6.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Peripheral Lung Tumor [Mean (Standard Deviation); unit: centimetre]
  Primary Tumor size - baseline | 1.70 (0.762)
  Metastatic Tumor size - baseline | 1.50 (0)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility to Perform Interstitial-Photodynamic Therapy (i-PDT) Into Tumor
Description: Number of times photodynamic therapy was delivered into the tumor using navigational bronchoscopy for each subject.
Time Frame: Day 3 post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
Participants
  One delivery of PDT into tumor | 3
  Two deliveries of PDT into tumor | 0
  Three deliveries of PDT into tumor | 1
  Four deliveries of PDT into tumor | 1

2. Primary Outcome: Adverse Events Incidence Indicating Safety of Navigational Bronchoscopy-interstitial-Photodynamic Therapy (i-PDT)
Description: The incidence of adverse events following navigational bronchoscopy-iPDT (interstitial-Photodynamic Therapy) will be presented as the primary safety indicator for this treatment.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
Participants
  Total number of participants with AEs | 5
  AE of Blood creatinine increased | 2
  AE of blood glucose increased | 2
  AE of heart rate increased | 2
  AE of laboratory test abnormal | 3
  AE of pulmonary function test abnormal | 3
  AE of respiratory rate increased | 2
  Erythema | 2
  Atelectasis | 2

3. Secondary Outcome: Tumor Response at 3 Months Post Photodynamic Therapy (PDT)
Description: From the start of treatment until 3 months post-treatment measured as per the Modified RECIST (Response Evaluation Criteria in Solid Tumors) Criteria
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
Participants
  Complete Response | 1
  Partial Response | 0
  Stable Response | 4
  Progression of Disease | 0
  Any response (Complete + Partial) | 1

4. Secondary Outcome: Tumor Response at Study Exit (6 Months) Post Photodynamic Therapy (PDT)
Description: From the start of treatment until 6 months post-treatment measured as per the Modified RECIST (Response Evaluation Criteria in Solid Tumors) Criteria
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
Participants
  Complete Response | 1
  Partial Response | 0
  Stable Response | 3
  Progression of Disease | 1
  Any response (Complete + Partial) | 1

5. Secondary Outcome: Performance Status on the Eastern Cooperative Oncology Group (ECOG) Score at Screening (Days -14 to -1). Baseline.
Description: Measured at screening to be the baseline measure. The Eastern Cooperative Oncology Group (ECOG) scores range from 0 to 5. The lowest values mean a better outcome: 0 is fully active with no performance restrictions; 1 is strenuous physical activity restricted but fully ambulatory and able to carry out light work; 2 is capable of all self-care but unable to carry out any work activities - up and about >50% of waking hours; 3 is capable of only limited self-care and confined to bed or chair >50% of waking hours; and 4 is completely disable, cannot carry out any self-care and totally confined to bed or chair.
Time Frame: up to day 0 (-14 to -1 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
Participants
  ECOG value of 0 | 1
  ECOG value of 1 | 2
  ECOG value of 2 | 2
  ECOG value of 3 | 0
  ECOG value of 4 | 0
  ECOG value of 5 | 0

6. Secondary Outcome: Performance Status on the Eastern Cooperative Oncology Group (ECOG) Score at Day 1 (Date of Photofrin Injection).
Description: Measured at Day 1 which is day of the photofrin injection. The Eastern Cooperative Oncology Group (ECOG) scores range from 0 to 5. The lowest values mean a better outcome: 0 is fully active with no performance restrictions; 1 is strenuous physical activity restricted but fully ambulatory and able to carry out light work; 2 is capable of all self-care but unable to carry out any work activities - up and about >50% of waking hours; 3 is capable of only limited self-care and confined to bed or chair >50% of waking hours; and 4 is completely disable, cannot carry out any self-care and totally confined to bed or chair.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
Participants
  ECOG value of 0 | 1
  ECOG value of 1 | 4
  ECOG value of 2 | 0
  ECOG value of 3 | 0
  ECOG value of 4 | 0
  ECOG value of 5 | 0

7. Secondary Outcome: Performance Status on the Eastern Cooperative Oncology Group (ECOG) Score at Day 3 (Day of Photodynamic Therapy)
Description: Measured at Day 3. The Eastern Cooperative Oncology Group (ECOG) scores range from 0 to 5. The lowest values mean a better outcome: 0 is fully active with no performance restrictions; 1 is strenuous physical activity restricted but fully ambulatory and able to carry out light work; 2 is capable of all self-care but unable to carry out any work activities - up and about >50% of waking hours; 3 is capable of only limited self-care and confined to bed or chair >50% of waking hours; and 4 is completely disable, cannot carry out any self-care and totally confined to bed or chair.
Time Frame: Day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 4
Participants
  ECOG value of 0 | 0
  ECOG value of 1 | 3
  ECOG value of 2 | 1
  ECOG value of 3 | 0
  ECOG value of 4 | 0
  ECOG value of 5 | 0

8. Secondary Outcome: Performance Status on the Eastern Cooperative Oncology Group (ECOG) Score at Day 30 (30 Days Post Photofrin Injection)
Description: as for outcome 7
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
Participants
  ECOG value of 0 | 1
  ECOG value of 1 | 2
  ECOG value of 2 | 2
  ECOG value of 3 | 0
  ECOG value of 4 | 0
  ECOG value of 5 | 0

9. Secondary Outcome: Performance Status on the Eastern Cooperative Oncology Group (ECOG) Score at 3 Months Post Photofrin Injection
Description: Measured at 3 months. The Eastern Cooperative Oncology Group (ECOG) scores range from 0 to 5. The lowest values mean a better outcome: 0 is fully active with no performance restrictions; 1 is strenuous physical activity restricted but fully ambulatory and able to carry out light work; 2 is capable of all self-care but unable to carry out any work activities - up and about >50% of waking hours; 3 is capable of only limited self-care and confined to bed or chair >50% of waking hours; and 4 is completely disable, cannot carry out any self-care and totally confined to bed or chair.
Time Frame: up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
Participants
  ECOG value of 0 | 2
  ECOG value of 1 | 2
  ECOG value of 2 | 1
  ECOG value of 3 | 0
  ECOG value of 4 | 0
  ECOG value of 5 | 0

10. Secondary Outcome: Performance Status on the Eastern Cooperative Oncology Group (ECOG) Score at 6 Months Post Photofrin Injection
Description: Measured at 6 months. The Eastern Cooperative Oncology Group (ECOG) scores range from 0 to 5. The lowest values mean a better outcome: 0 is fully active with no performance restrictions; 1 is strenuous physical activity restricted but fully ambulatory and able to carry out light work; 2 is capable of all self-care but unable to carry out any work activities - up and about >50% of waking hours; 3 is capable of only limited self-care and confined to bed or chair >50% of waking hours; and 4 is completely disable, cannot carry out any self-care and totally confined to bed or chair.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
Participants
  ECOG value of 0 | 3
  ECOG value of 1 | 1
  ECOG value of 2 | 1
  ECOG value of 3 | 0
  ECOG value of 4 | 0
  ECOG value of 5 | 0

11. Secondary Outcome: Short Form Health Survey (SF-36) Score at Baseline
Description: The Short-Form Health Survey (SF-36) scores range from 0 to 100, with higher scores indicating better health status. SF-36 evaluates 9 dimensions of Health: physical function, role limitations due to physical health problems, body pain, general health, vitality, social functioning, role limitations due to emotional problems domain, and mental health. Summary is provided in the form of physical component score (PCS) and mental component score (MCS) for each of the timepoints.
Time Frame: Baseline
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
score on a scale
  Physical Component Score (PCS) | 49.27 (6.71)
  Mental Component Score | 29.47 (3.13)

12. Secondary Outcome: Short-Form Health Survey (SF-36) Score at Follow-up Visit at 3 Months.
Description: as for outcome 11
Time Frame: up to 3 months
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
score on a scale
  Physical Component Score (PCS) | 46.83 (5.60)
  Mental Component Score (MCS) | 30.04 (8.64)

13. Secondary Outcome: Short-Form Health Survey (SF-36) Score at Study Exit (6 Month Visit)
Description: as for outcome 11
Time Frame: Up to 6 months
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
score on a scale
  Physical Component Score (PCS) | 48.33 (7.45)
  Mental Component Score (MCS) | 31.90 (9.61)

14. Secondary Outcome: Health-related Quality of Life on the 4- and 7-point European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire 30 Item (QLQ-C30): Baseline
Description: Baseline score of EORTC QLQ-C30 which is a multi-dimensional Health Related Quality of Life measure designed for use in lung cancer patients. Includes 5 functional measures (physical, role, emotional, social, cognitive), 8 symptoms (fatigue, pain, nausea/vomiting, appetite loss, constipation, diarrhea, insomnia, dyspnea) and global health status and financial impact. Most items use 4-item scale from "not at all" to "very much". Raw scores are transformed to 0-100 scale with higher scores representing better functioning/Quality of Life and greater symptom burden.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
score on a scale
  Global Health Status | 55.0 (28.62)
  Physical Functioning | 73.34 (10.55)
  Role Functioning | 60.02 (30.27)
  Emotional Functioning | 80.0 (17.29)
  Cognitive Functioning | 76.66 (18.99)
  Social Functioning | 70.0 (41.50)
  Fatigue | 24.44 (25.35)
  Nausea and Vomiting | 3.34 (7.47)
  Pain | 43.34 (27.91)
  Dyspnoea | 53.32 (44.73)
  Insomnia | 20.0 (29.82)
  Appetite Loss | 26.64 (14.89)
  Constipation | 6.66 (14.89)
  Diarrhoea | 6.66 (14.89)
  Financial Difficulties | 46.66 (50.56)

15. Secondary Outcome: Health-related Quality of Life on the 4- and 7-point European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire 30 Item (QLQ-C30): Follow-up 3 Months
Description: 3 month score of EORTC QLQ-C30 which is a multi-dimensional Health Related Quality of Life measure designed for use in lung cancer patients. Includes 5 functional measures (physical, role, emotional, social, cognitive), 8 symptoms (fatigue, pain, nausea/vomiting, appetite loss, constipation, diarrhea, insomnia, dyspnea) and global health status and financial impact. Most items use 4-item scale from "not at all" to "very much". Raw scores are transformed to 0-100 scale with higher scores representing better functioning/Quality of Life and greater symptom burden.
Time Frame: up to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
score on a scale
  Global Health Status | 70.0 (17.29)
  Physical Functioning | 68.0 (20.76)
  Role Functioning | 63.34 (24.73)
  Emotional Functioning | 80.02 (12.63)
  Cognitive Functioning | 73.34 (18.99)
  Social Functioning | 80.0 (21.72)
  Fatigue | 28.86 (12.66)
  Nausea and Vomiting | 6.66 (14.89)
  Pain | 30.0 (29.82)
  Dyspnoea | 60.0 (27.91)
  Insomnia | 13.32 (18.24)
  Appetite Loss | 26.66 (27.90)
  Constipation | 20.0 (29.82)
  Diarrhoea | 26.66 (27.90)
  Financial Difficulties | 33.32 (40.83)

16. Secondary Outcome: Health-related Quality of Life on the 4- and 7-point European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire 30 Item (QLQ-C30): 6 Months
Description: 6 month score of EORTC QLQ-C30 which is a multi-dimensional Health Related Quality of Life measure designed for use in lung cancer patients. Includes 5 functional measures (physical, role, emotional, social, cognitive), 8 symptoms (fatigue, pain, nausea/vomiting, appetite loss, constipation, diarrhea, insomnia, dyspnea) and global health status and financial impact. Most items use 4-item scale from "not at all" to "very much". Raw scores are transformed to 0-100 scale with higher scores representing better functioning/Quality of Life and greater symptom burden.
Time Frame: Up to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
score on a scale
  Global Health Status | 71.66 (20.07)
  Physical Functioning | 58.66 (22.80)
  Role Functioning | 66.68 (35.34)
  Emotional Functioning | 75.0 (22.03)
  Cognitive Functioning | 76.66 (9.09)
  Social Functioning | 76.68 (14.89)
  Fatigue | 28.88 (21.67)
  Nausea and Vomiting | 0 (0)
  Pain | 36.66 (13.94)
  Dyspnoea | 53.34 (38.02)
  Insomnia | 13.32 (18.24)
  Appetite Loss | 19.98 (18.24)
  Constipation | 13.32 (18.24)
  Diarrhoea | 13.32 (18.24)
  Financial Difficulties | 33.32 (40.83)

17. Secondary Outcome: Health-related Quality of Life on the 4- Point European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire for Lung Cancer 13 Item (QLQ-LC13): Baseline Score
Description: Baseline measure for EORTC QLQ-LC13 which is a 13-item lung cancer-specific questionnaire module. It is used in conjunction with the QLQ-C30. It is comprised of multi-item and single-item measures of lung cancer associated symptoms (coughing, hemoptysis, dyspnea, pain) and side effects from conventional chem-and radiotherapy (alopecia, neuropathy, sore mouth, dysphagia). For these symptom-oriented scales, a higher score means more severe symptoms. The scale is from 1 (not at all) to 4 (very much). The scoring (as reported here) is from 0 to 100 with the higher score meaning a more severe symptom.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
score on a scale
  Dyspnea | 39.98 (24.36)
  Coughing | 33.32 (23.58)
  Haemoptysis | 6.66 (14.89)
  Sore Mouth | 6.66 (14.89)
  Dysphagia | 20.0 (29.82)
  Peripheral Neuropathy | 19.98 (18.24)
  Alopecia | 33.34 (47.15)
  Pain in Chest | 6.66 (14.89)
  Pain in Arm or Shoulder | 19.98 (18.24)
  Pain in Other Parts | 40.0 (27.91)

18. Secondary Outcome: Health-related Quality of Life on the 4- Point European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire for Lung Cancer 13 Item (QLQ-LC13): Follow-up 3 Month Score
Description: 3-Month measure for EORTC QLQ-LC13 which is a 13-item lung cancer-specific questionnaire module. It is used in conjunction with the QLQ-C30. It is comprised of multi-item and single-item measures of lung cancer associated symptoms (coughing, hemoptysis, dyspnea, pain) and side effects from conventional chem-and radiotherapy (alopecia, neuropathy, sore mouth, dysphagia). For these symptom-oriented scales, a higher score means more severe symptoms. The scale is from 1 (not at all) to 4 (very much). The scoring (as reported here) is from 0 to 100 with the higher score meaning a more severe symptom.
Time Frame: up to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
score on a scale
  Dyspnea | 40.0 (24.37)
  Coughing | 26.64 (14.89)
  Haemoptysis | 0 (0)
  Sore Mouth | 13.32 (18.24)
  Dysphagia | 13.32 (18.24)
  Peripheral Neuropathy | 19.98 (18.24)
  Alopecia | 26.66 (43.46)
  Pain in Chest | 6.66 (14.89)
  Pain in Arm or Shoulder | 19.98 (18.24)
  Pain in Other Parts | 66.66 (33.35)

19. Secondary Outcome: Health-related Quality of Life on the 4- Point European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire for Lung Cancer 13 Item (QLQ-LC13): Study Exit (6 Months) Score
Description: 6-Month measure for EORTC QLQ-LC13 which is a 13-item lung cancer-specific questionnaire module. It is used in conjunction with the QLQ-C30. It is comprised of multi-item and single-item measures of lung cancer associated symptoms (coughing, hemoptysis, dyspnea, pain) and side effects from conventional chem-and radiotherapy (alopecia, neuropathy, sore mouth, dysphagia). For these symptom-oriented scales, a higher score means more severe symptoms. The scale is from 1 (not at all) to 4 (very much). The scoring (as reported here) is from 0 to 100 with the higher score meaning a more severe symptom.
Time Frame: Up to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
score on a scale
  Dyspnea | 40.0 (30.04)
  Coughing | 39.98 (14.94)
  Haemoptysis | 0 (0)
  Sore Mouth | 6.66 (14.89)
  Dysphagia | 23.66 (43.46)
  Peripheral Neuropathy | 33.32 (23.58)
  Alopecia | 26.66 (43.46)
  Pain in Chest | 6.66 (14.89)
  Pain in Arm or Shoulder | 40.0 (27.91)
  Pain in Other Parts | 26.66 (27.9)

20. Secondary Outcome: Number of Participants With Indicated Adverse Events
Description: Adverse events (AEs) noted by number of participants with at least one event. An AE was defined as any untoward medical occurrence in a subject during the course of the study, regardless of causal relationship. AEs were coded using MedDRA Version 21.1
Time Frame: Up to 6 months post-treatment
Measure: Number; unit: Participants with at least one event
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
Participants with at least one event
  Porphyria Grade 2 | 1
  Eye oedema grade 1 | 1
  Dysphagia grade 1 | 1
  Asthenia Grade 1 | 1
  Oedema peripheral grade 1 | 1
  Fall grade 1 | 1
  Trunk injury grade 1 | 1
  Blood pressure increased grade 1 | 2
  Breath sounds abnormal grade 1 | 1
  Carbon monoxide diffusing capacity decreased gr. 1 | 1
  Creatinine renal clearance abnormal gr. 1 | 1
  Heart rate increased grade 1 | 1
  Oxygen saturation decreased grade 1 | 1
  Pulmonary function test abnormal grade 1 | 2
  Respiratory rate increased grade 1 | 2
  Back pain grade 1 | 1
  Atelectasis grade 1 | 2
  Pleural effusion grade 1 | 1
  Dermatitis grade 1 | 1
  Erythema grade 1 | 1
  Erythema grade 2 | 1
  Hyperkeratosis grade 1 | 1
  Photosensitivity reaction grade 2 | 1
  Pruritus grade 1 | 1
  Rash grade 1 | 1
  Skin exfoliation grade 1 | 1
  Flushing grade 1 | 1

21. Secondary Outcome: Number of Subjects With at Least One Serious Adverse Event
Description: The number of subjects with at least one serious adverse event are listed.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
Participants | 0

22. Secondary Outcome: Safety: Physical Examination Summaries for Each Subject
Description: Safety evaluation will include the physical examinations summary of non-normal findings for each subject.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
Participants
  Abnormal eyes at 3 month follow-up | 1
  Abnormal nose, throat, ears and mouth at day 3 | 1
  Abnormal skin at screening | 2
  Abnormal skin at Day 1 | 2
  Abnormal skin at Day 3 | 2
  Abnormal skin at Day 5 | 1
  Abnormal skin at day 10 | 4
  Abnormal skin at day 30 | 3
  Abnormal skin at 3 months | 1
  Abnormal skin at 6 months | 1
  Abnormal respiratory at screening | 1
  Abnormal respiratory at day 1 | 2
  Abnormal respiratory at day 3 | 2
  Abnormal respiratory at day 5 | 2
  Abnormal respiratory at day 10 | 1
  Abnormal respiratory at day 30 | 2
  Abnormal respiratory at 3 months | 2
  Abnormal respiratory at 6 months | 1
  Abnormal abdomen/Gastrointestinal Day 1 | 1
  Abnormal abdomen/Gastrointestinal 3 months | 1
  Abnormal neurological at screening | 1

23. Secondary Outcome: Safety: Number of Participants With Indicated Vital Sign Summaries
Description: Safety evaluation included vital sign summary for each subject. Vital signs included pulse, blood pressure, temperature and respiration rate. Only clinically relevant results, as per the investigator judgement, are included. These would be vital signs that are out of the normal range but could be considered outside enough to be clinically relevant to the subject's health.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
Participants
  Blood pressure increased study day 180 grade 1 | 1
  Respiratory rate increased study day 180 grade 1 | 1
  Respiratory rate increased day 3 grade 1 | 1
  Heart rate increased day 5 grade 1 | 1
  Blood pressure increased day 31 grade 1 | 1

24. Secondary Outcome: Safety: Number of Participants With Indicated Changes to Pulmonary Function Tests (PFTs) Related to Treatment Emergent Adverse Events
Description: The treatment emergent adverse events related to PFTs are noted. Pulmonary function test measurements were: Diffusion Capacity of Lung for Carbon Monoxide (%), Expiratory Reserve Volume (mL), Forced Vital Capacity (mL), Forced Expiratory Volume in 1 second (mL), Forced Expiratory Flow 25% to 75% (L/min), Functional Residual Capacity (mL), Maximum Voluntary Ventilation (L/min), Residual Volume (mL), Peak Expiratory Flow (L/min), Slow Vital Capacity (mL), Total Lung Capacity (mL)
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
Participants
  Carbon Monoxide Diffusing Capacity down Day 92 g.1 | 1
  Expiratory Reserve Volume decreased Day 92 grade 1 | 1
  Forced Expiratory Volume abnormal Day 92 grade 1 | 1
  Forced Vital Capacity Abnormal Day 92 Grade 1 | 1
  Carbon Monoxide Diffusing Capacity down 3 mos. g.1 | 1
  Expiratory Reserve Volume decreased 3 mos. grade 1 | 1
  Forced Expiratory Volume abnormal 3 mos. grade 1 | 1
  Forced Vital Capacity Abnormal 3 mos. Grade 1 | 1
  Oxygen Saturation decreased Day 5 grade 1 | 1

25. Secondary Outcome: Safety: Laboratory Test Summaries for Each Subject
Description: Safety evaluation includes laboratory tests summarized for each subject with any abnormal lab results considered an Adverse Event to be listed. The investigators commented on any laboratory value outside the normal reference range. If the value was judged to be an Adverse Event, it is listed. The values analysed were: Hematology (Hemoglobin, Hematocrit, White Blood Cell, Red Blood Cell, Platelet Count, Prothrombin Time) and Chemistry (Glucose (random), Blood Urea Nitrogen, Electrolytes (sodium, potassium, chloride), Creatinine, Alkaline Phosphatase, Aspartate Aminotransferase, Alanine Aminotransferase, Total Bilirubin, Albumin, Total Protein)
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
Participants
  High post-baseline alkaline phosphatase | 2
  High Alkaline Phosphatase value from baseline | 1
  High post-baseline alanine transaminase | 1
  High aspartate transaminase from baseline | 1
  High creatinine levels from baseline | 2
  High post-baseline glucose levels | 1
  High glucose levels from baseline | 3
  High urea nitrogen post baseline | 2
  High protein post baseline | 1
  High post baseline hematocrit | 1
  Low hematocrit values from baseline | 2
  Low erythrocyte count from baseline | 2
  High erythrocyte count from baseline | 1
  High leukocyte count from baseline | 1
  High leukocyte at baseline & then normal post base | 1

26. Other Pre Specified Outcome: Immunology Markers Concentrations Were Examined as an Exploratory Endpoint. The Change From Baseline Was Reported.
Description: Distribution of lymphocyte subsets from peripheral blood was determined by flow cytometry. Flow cytometry is a laser-based technique used to detect and measure physical and chemical characteristics of a population of cells or particles. It allows simultaneous multi-parameter analysis of single cells.
  The selected markers of interest, representative of the broader markers were: Total Thymus-cells (T-Cells), Cluster of Differentiation 4 (CD4) T cell subsets, and Cluster of Differentiation 9 (CD8) T cell subset, CD4 T Regulatory (T Reg) cells, Natural Killer Cells, Activated T cells, Myeloid-Derived Suppressor Cells (MSCDs), Monocytes. The Percent Gated and Absolute counts were analysed for each marker. Gating allows the analysis to be restricted to a specific size of cells (e.g. lymphocytes) to allow a more specific analysis. Absolute counting quantifies the total number of cells. It is recommended to look at both values to get the full picture.
Time Frame: Baseline, 10 days post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
Participants
  CD45+ cells Percent gated increased | 2
  CD45+ cells Percent gated decreased | 3
  CD45+ cells Absolute Count increased | 2
  CD45+ cells Absolute Count decreased | 3
  Helper T cells Percent Gated Increased | 3
  Helper T cells Percent Gated Decreased | 1
  Helper T cells Percent Gated stayed the same | 1
  Helper T cells Absolute counts Increased | 1
  Helper T cells Absolute counts Decreased | 4
  CD3+, CD4+ T cells Percent Gated increased | 4
  CD3+, CD4+ T cells Percent Gated decreased | 1
  CD3+, CD4+ T cells Absolute Counts increased | 1
  CD3+, CD4+ T cells Absolute Counts decreased | 4
  T Reg Cells Percent Gated increased | 3
  T Reg Cells Percent Gated decreased | 1
  T Reg Cells Percent Gated similar | 1
  T Reg Cells Absolute Counts increased | 1
  T Reg Cells Absolute Counts decreased | 4
  Cytotoxic T Cells Percent Gated increased | 1
  Cytotoxic T Cells Percent Gated decreased | 3
  Cytotoxic T Cells Percent Gated similar | 1
  Cytotoxic T Cells Absolute Counts increased | 1
  Cytotoxic T Cells Absolute Counts decreased | 4
  Natural Killer Cells Percent Gated increased | 2
  Natural Killer Cells Percent Gated decreased | 1
  Natural Killer Cells Percent Gated Not Done | 2
  Natural Killer Cells Absolute Counts increased | 2
  Natural Killer Cells Absolute Counts decreased | 1
  atural Killer Cells Absolute Counts Not Done | 2
  Activated T Cells Percent Gated Increased | 3
  Activated T Cells Percent Gated Decreased | 2
  Activated T Cells Absolute Counts Increased | 2
  Activated T Cells Absolute Counts Decreased | 3
  TH17 Cytokines Percent Gated Increased | 1
  TH17 Cytokines Percent Gated Decreased | 2
  TH17 Cytokines Percent Gated Not Done | 2
  TH17 Cytokines Absolute Counts Increased | 2
  TH17 Cytokines Absolute Counts Decreased | 3
  Monocytic MDSCs Percent Gated Increased | 3
  Monocytic MDSCs Percent Gated Decreased | 2
  Monocytic MDSCs Absolute Counts Increased | 3
  Monocytic MDSCs Absolute Counts Decreased | 2
  Granulocytic MDSCs Percent Gated Increased | 3
  Granulocytic MDSCs Percent Gated Decreased | 2
  Granulocytic MDSCs Absolute Counts Increased | 3
  Granulocytic MDSCs Absolute Counts Decreased | 2
  Monocytes Percent Gated Increased | 4
  Monocytes Percent Gated Decreased | 1
  Monocytes Absolute Counts Increased | 3
  Monocytes Absolute Counts Decreased | 2

27. Other Pre Specified Outcome: Skin Photosensitivity as a Adverse Event of Special Interest: Participants With Event
Description: Adverse Event of special interest was Skin Photosensitivity. Skin photosensitivity was examined because all subjects who receive Photofrin are photosensitive and must observe precautions to avoid exposure of eyes and skin to direct sunlight or bright indoor lights for 30 days or longer. Changes in skin will be assessed by grade of erythema, edema and blistering and will be tabulated by Common Terminology Criteria for Adverse Events (CTCAE) grade in the dermatology/skin category.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy-Photofrin
Number analyzed (Participants) | 5
Participants
  Erythema Grade 1 Events; related | 1
  Erythema Grade 2 Events; related | 1
  Photosensitivity Reaction Grade 2; related | 1
  Rash grade 1; related | 1
  Skin Exfoliation grade 1; related | 1
  Flushing grade 1; related | 1

ADVERSE EVENTS:
Time Frame: 6 months for each subject. The study was conducted over a period of 1 year and 5 months in total (29Nov2017 to 12Apr2019)
Arm/Group | Photodynamic Therapy-Photofrin
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Photodynamic Therapy-Photofrin (N=5)
Porphyria (Congenital, familial and genetic disorders) | 1 (1)
Eye Oedema (Eye disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Peripheral Oedema (General disorders) | 1 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Trunk Injury (Injury, poisoning and procedural complications) | 1 (1)
Blood Creatinine Increased (Investigations) | 2 (3)
Blood Glucose Increased (Investigations) | 2 (3)
Blood Pressure Abnormal (Investigations) | 1 (1)
Blood Pressure Decreased (Investigations) | 1 (1)
Blood Pressure Diastolic Increased (Investigations) | 1 (2)
Blood Pressure Increased (Investigations) | 2 (4)
Blood Pressure Systolic Increased (Investigations) | 1 (4)
Breath Sounds Abnormal (Investigations) | 1 (2)
Carbon Monoxide diffusing capacity decreased (Investigations) | 2 (3)
Chest X-Ray Abnormal (Investigations) | 1 (2)
Creatinine Renal Clearance Abnormal (Investigations) | 1 (1)
Expiratory Reserve Volume decreased (Investigations) | 1 (1)
Forced Expiratory Volume abnormal (Investigations) | 2 (3)
Forced Vital Capacity abnormal (Investigations) | 2 (2)
Haematocrit decreased (Investigations) | 1 (3)
Haemoglobin decreased (Investigations) | 1 (3)
Heart Rate decreased (Investigations) | 1 (2)
Heart Rate increased (Investigations) | 2 (2)
Laboratory test abnormal (Investigations) | 4 (7)
Oxygen Consumption decreased (Investigations) | 1 (5)
Oxygen Saturation decreased (Investigations) | 1 (2)
Pulmonary Function Test abnormal (Investigations) | 3 (5)
Red Blood Cell Count Decreased (Investigations) | 2 (7)
Respiratory Rate increased (Investigations) | 2 (4)
White Blood Cell Count abnormal (Investigations) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (11)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Electrocardiogram abnormal (Investigations) | 1 (1)
Blood Albumin increased (Investigations) | 1 (1)
Blood Urea increased (Investigations) | 1 (1)
Glomerular Filtration Rate abnormal (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination of the study lead to small numbers of subject being analysed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT02916745/Prot_SAP_001.pdf